CLINICAL TRIAL: NCT07200700
Title: Assessing Knee Laxity and Inter-rater Reliability of the GNRB Arthrometer a Clinical Study of Patients With Anterior Cruciate Ligament Injuries Before and After Reconstruction
Brief Title: Inter-rater Reliability of the GNRB Arthrometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Ninni Sernert, Professor, Research director, Vastra Gotaland Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dnr 2020-02062
Record Dates: First submitted 2025-09-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior cruciate ligament reconstruction, arthrometers, GNRB, KT1000, knee laxity

STUDY DESIGN:
Intervention Model Description: Inter-reliablility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GNRB arthrometer (Other): Reliability testing GNRB arthrometer between two examinors
  Interventions: Diagnostic Test: Knee laxity arthrometer

INTERVENTIONS:
Diagnostic Test: Knee laxity arthrometer — Inter-reliability analysis of the GNRB arthrometer between two examinors compared to standard KT 1000 arthrometer

SUMMARY:
Although clinical examination is commonly used to diagnose an anterior cruciate ligament (ACL) injury, the method is subjective. For many years, the arthrometer KT1000 has been used to verify clinical results, mostly due to its simplicity. While the KT1000 is no longer available for purchase, other arthrometers have been introduced, one being the Genoroub (GNRB). The latter has several automatic steps, has been marketed to have a higher reproducibility, and able to detect partial tears.

While the KT1000 and GNRB have previously been compared in several studies, it's mostly been compared in healthy subjects. The current study aim to analyse the results in a clinical environment on injured objects and compare the results both before and after ACL reconstruction. The main hypothesis was that the GNRB offers high inter-rater reliability between two examinors and can replace the KT1000 in the everyday clinical setting.

Methods Consecutively, 20 patients > 18 years of age, 12 men and 8 women, with an ACL injury scheduled for surgical reconstruction, were included. All patients were screened between August 2020-2021 at the NU Hospital Group in Trollhattan, Sweden. To be eligible, the patients had to present with a first time ACL injury verified by clinical examination with or without an magnetic resonance imaging, a healthy contralateral knee and to not have sustained multi-ligament injuries to the knee. Minor collateral ligament injuries and meniscal and cartilage injuries were included.

All patients received both spoken and written information before signing an informed consent. The study was approved by the Swedish ethical committee.

All patients were examined both pre- and postoperatively, in accordance with local standard protocol, including range of motion, knee laxity measurements (manual Lachman test, pivot shift test) The participants were examined starting with the healthy/uninjured knee. Who of the two examinors started the testing was randomly decided, however alternated at the follow-up. Clinical examination and KT1000 testing were only performed by examiner 2, given the need for experience with the KT1000 for accurate results.

Statistically, a side-to-side difference (SSD) of 3 mm was set to indicate ACL injury according to general concensus. For the dichotomous values, an SSD of ≥3 mm was considered a yes to ACL injury and <3mm a no, respectively, for both the GNRB and the KT1000.

A power analysis was performed estimating a difference of 1 mm between examiners with an SD of 1 mm, resulting in 17 patients needed to reach a power of 80% with a significance level of 0.05.

As for the inter-rater reliability, the intra-correlation coefficient (ICC) was calculated and considered poor (<0.5), moderate (0.5-0.75), good (0.75-0.9) or excellent (>0.9).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Patients under 18 years of age, and those having had previous surgery to any knee, posterior cruciate ligament (PCL) injury or more severe concomitant injuries to the meniscus and collateral ligaments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Identifying anterior knee translation in patients with anterior cruciate ligament injury before and after reconstruction compared to the contralateral non-injured knee | Primary measurement pre operative, secondary measurement 6-12 months after reconstruction
  Measuring anterior knee translation in both injured and non injured knee before and after reconstruction using two different devices; GNRB and KT 1000 arthrometer

CONTACTS AND LOCATIONS:
Locations (1):
- NU Hospital Group, Trollhättan, Europe, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As the study is a part of future thesis data will be available in this publication
Supporting Information: ICF
Time Frame: At earliest 2027
Access Criteria: The future thesis will be available both as a printed book and in digital form
URL: https://isp.gu.se/isp/externalLogin